CLINICAL TRIAL: NCT01377701
Title: The Predictive Factors of Vision Recovery in Patients With Pituitary Tumor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Yao Zhao, Huashan Hospital
Other Study IDs: KY2010-259
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Pituitary Adenomas
Keywords: pituitary adenomas; recovery of vision; trans-sphenoidal surgery
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pituitary adenomas can cause compression of optic nerves and chiasm, which will lead to damage of vision. This study aims to evaluate the predictive factors for recovery of vision in patients with pituitary adenomas following trans-sphenoidal surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* patients with pituitary adenomas, loss of visual field
* patients receive trans-sphenoidal surgery

Exclusion Criteria:

* visual damage caused by other diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pituitary adenomas at Huashan Hospital will be screened. Patients with loss of visual field and receive trans-sphenoidal surgery will be included.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhao, M.D., Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China